CLINICAL TRIAL: NCT04835259
Title: Efficacy of a Combination of Topical Antioxidants in Tretment of Photoaged Skin:A Randomized Controlled Trial
Brief Title: Efficacy of Topical Antioxidants in Tretment of Photoaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, esraa ismail, assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-21-01-10
Record Dates: First submitted 2021-01-19; First posted 2021-04-08 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Photoaging
Keywords: topical antioxidants; photoaged skin
MeSH Terms: interventions — Retinoids; dexpanthenol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1(treatment group) (Active Comparator): Topical application of a cream of a combination of antioxidants once daily at night for 6 months Name: Selenium ACE cream (Interpharma UK company, Egypt)
  Ingredients:
  Selenium (Selenium amino acid chelate) 0.5% Vitamin C (Sodium ascorbyl phosphate - stay C) %1 Vitamin E (Tocopheryl acetate) % 0.5 Vitamin A (Retinyl palmitate) %1 Emulsifiers ( Ceteareth 20 , Glycerol monostearate , Cetyl alcohol) Emollient(Caprylic capric triglycerides)
  Interventions: Drug: Selenium Amino Acid Chelate (Selenium ACE cream)
- Group 2 (positive control) (Active Comparator): Topical application of a retinoid (tretinoin 0.05%) cream once daily at night for 6 months (Acretin 0.05% cream Jamjoom pharmaceuticals, Egypt)
  Interventions: Drug: Selenium Amino Acid Chelate (Selenium ACE cream)
- Group 3 (Negative control) (Placebo Comparator): Topical application of a panthenol cream once daily at night for 6 months (panthenol 2% cream, El Nile company, Egypt)
  Interventions: Drug: Selenium Amino Acid Chelate (Selenium ACE cream)

INTERVENTIONS:
Drug: Selenium Amino Acid Chelate (Selenium ACE cream) — application of a topical agent over the whole face for 6 months
  Other Names: topical retinoid (Acretin 0.05% cream); topical panthenol (Panthenol cream)

SUMMARY:
This randomized controlled trial study aims at investigating the efficacy and safety of topical antioxidants in treatment of a cohort of non-elderly volunteers with photoaged skin.

DETAILED DESCRIPTION:
•Sample size calculation: The sample size was assessed prospectively using Openepi version 3.01 to provide a 80% power to detect a 40-50% difference before and after treatment using either topical antioxidants or retinoids with a significance level of 0.05 (based on the results of a previous clinical trial). Assuming 10% dropout, 30 patients will be recruited in each treatment group.

•Statistical analysis: Data will be collected and recorded on excel data sheet. Data will be tested for normality. Quantitative data will be represented as mean and standard deviation, or median and interquartile range. Qualitative data will be presented as number and percentage. The relevant statistical method will be used for comparison. P value will be considered statistically significant if it is less than 0.05

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers < 50 years old
* Clinical and dermoscopic features of photoaging.

Exclusion Criteria:

* Genodermatoses associated with photosensitivity.
* Treatment by medications affecting skin aging (eg, topical and systemic retinoids) in the last 6 months prior to enrollment.
* Any recent cosmetic procedures.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
change in Dermoscopy photoaging scale | assesed every month for 6 months
  Dermoscopy photoaging scale (DPAS) is a reliable and valid diagnostic tool that can evaluate photoaged skin quantitatively by the help of objective criteria. It can be used to evaluate the effect of preventive and therapeutic applications for skin aging.

CONTACTS AND LOCATIONS:
Overall Officials: esraa ismail, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No